CLINICAL TRIAL: NCT06036342
Title: Atrial Fibrillation Screening With MobiCARE in Subjects With Health Care Examination
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Other Study IDs: AF-CARE
Record Dates: First submitted 2023-03-20; First posted 2023-09-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MobiCARE test — 7-days continuous electrocardiography monitoring using MobiCARE device

SUMMARY:
This study aimed to detect and diagnose atrial fibrillation early by conducting a screening test for atrial fibrillation using a continuous electrocardiography monitoring device for those who have undergone a health screening examination.

Early detection through atrial fibrillation screening tests in high-risk patients with stroke is intended to prevent stroke by starting stroke prevention treatment early. It is intended to detect asymptomatic atrial fibrillation patients early through examination and ultimately improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 65 years or older who have at least one stroke risk factor*
2. Subjects aged 19 years to <65 years who have two or more stroke risk factors.
3. Subjects aged 75 years or older

   * Stroke risk factors: heart failure, hypertension, diabetes, vascular disease, women, stroke/systemic embolism/transient ischemic attack (although stroke/systemic embolism/transient ischemic attack among stroke risk factors is considered to have two risk factors)
   * Heart failure: a history of heart failure diagnosis or a history of current heart failure treatment.
   * Hypertension, Diabetes: Diagnostic History
   * Vascular diseases: Significant coronal atherosclerosis (when 70% or more of the computed tomography or coronary angiography is present or coronary intervention is performed), 50% or more of the carotid artery disease, peripheral vascular disease, history of myocardial infarction, and aortic plaques

Exclusion Criteria:

1. Subjects diagnosed with atrial fibrillation in the past
2. Subjects aged under 19 years and other vulnerable research subjects
3. Subjects who have patch-type adhesive allergies/atopy dermatitis/ urticaria/skin rash/hives that are difficult to apply patches continuously
4. Subjects who have a structural abnormality in the thorax and is difficult to attach the device.
5. Subjects who have cardiac implantable electronic device (pacemaker, implantable cardioverter-defibrillator, implantable loop recorder, or cardiac resynchronized therapy-pacemaker or defibrillator)
6. Subjects requiring immediate ECG analysis or ECG monitoring through hospitalization due to arrhythmia that can be life-threatening
7. Subjects who are deemed inappropriate to participate in the research as judged by the researcher for other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those who have undergone a health screening examination.
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation detection rate | 1 year
  Atrial fibrillation detection rate at 1-year follow-up time

SECONDARY OUTCOMES:
The detection rate of atrial fibrillation | up to 7 days
  The detection rate of atrial fibrillation
The burden of atrial fibrillation. | up to 7 days
  The burden of atrial fibrillation.
The detection rate of other arrhythmias | up to 7 days
  The detection rate of other arrhythmias in addition to atrial fibrillation
The rate of initiation of antiarrhythmic and anticoagulant therapy, and the rate of receiving treatment related to rhythm control | 1 year
  The rate of initiation of antiarrhythmic and anticoagulant therapy, and the rate of receiving treatment related to rhythm control at 1-year follow-up time
Clinical outcome during 1-year follow-up. | 1 year
  stroke, transient ischemic attack, systemic embolism, admission for heart failure, admission for atrial fibrillation manage/control, cardiac arrest, cardiovascular death, and all-cause death
Evaluation of the convenience of wearing and using the Mobicare device | up to 1 month
  Questionnaire about convenience of wearing and using the Mobicare device
  1. Did you feel uncomfortable going about your daily routine, and mainly when?
  2. If you felt uncomfortable, what were your main concerns?
  3. If your skin itches or breaks out in a rash during use, how long has it been since you've been wearing it?
  4. How much discomfort did you experience due to foreign body sensation, skin problems, etc.?
  5. Has your device ever been dropped while in use? If so, when did it happen?
  6. Were there any challenges in reattaching the device, and if so, what were they?
  7. How often have you taken your device off and put it back on?
  8. How long do you think you can run the test without too much inconvenience?

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No